CLINICAL TRIAL: NCT06562010
Title: Evaluating the Efficacy of Culturally Adapted Internet-Delivered Cognitive Therapy for Social Anxiety Disorder (iCT-SAD) in Pakistan
Brief Title: Evaluating the Efficacy of Culturally Adapted iCT-SAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: Green International University (Other)
Responsible Party: Principal Investigator, Arshed Muhammad, PhD studentship, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: UIMT
Record Dates: First submitted 2024-08-17; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Social Anxiety; ICT

STUDY DESIGN:
Intervention Model Description: It is a two-arm 1:1 randomized control trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, care providers and outcome assessors will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention arm will receive a Pakistani version of Internet-delivered Cognitive Therapy for Social Anxiety Disorder (iCT-SAD), assessing its effectiveness in reducing social anxiety symptoms among Pakistani individuals. This will involve culturally tailored online therapy modules, therapist support, and regular progress assessments.
  Interventions: Behavioral: iCT-SAD-PK
- Control (No Intervention): The control arm will receive no intervention except usual care.

INTERVENTIONS:
Behavioral: iCT-SAD-PK — The intervention arm will receive a Pakistani version of Internet-delivered Cognitive Therapy for Social Anxiety Disorder (iCT-SAD), assessing its effectiveness in reducing social anxiety symptoms among Pakistani individuals. This will involve culturally tailored online therapy modules, therapist support, and regular progress assessments.
  Arms: Intervention group

SUMMARY:
The study will adapt and implement a Pakistani version of Internet-delivered Cognitive Therapy for Social Anxiety Disorder (iCT-SAD), assessing its effectiveness in reducing social anxiety symptoms among Pakistani individuals.

DETAILED DESCRIPTION:
The study will adapt and implement a Pakistani version of Internet-delivered Cognitive Therapy for Social Anxiety Disorder (iCT-SAD), assessing its effectiveness in reducing social anxiety symptoms among Pakistani individuals. This randomized controlled trial will involve culturally tailored online therapy modules, therapist support, and regular progress assessments. The goal is to evaluate the efficacy of iCT-SAD in a Pakistani context, comparing outcomes to a control group. The primary outcome measure is the self-report Liebowitz Social Anxiety Scale, and secondary outcomes include other measures of social anxiety symptoms and processes, general mood and functioning, and response to treatment

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of SAD based on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* Aged 18-75 years
* Regular, access to an appropriate internet device
* Resident of Pakistan and can write and speak Urdu
* Participants not currently undertaking other structured psychological therapy during the trial

Exclusion Criteria:

* Current psychosis, bipolar disorder, antisocial personality disorder, or alcohol/substance use disorder
* Active suicidal ideation with intent or plan
* Previously received CT or cognitive behavioral therapy for SAD

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2024-08-25 (Estimated); Primary Completion 2025-02-05 (Estimated); Study Completion 2025-03-25 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is change in Social Anxiety score (LSAS) | 6-months from baseline
  The primary outcome will be measured by Liebowitz Social Anxiety Scale. The 24 items are first rated on a Likert Scale from 0 to 3 on fear felt during the situations, and then the same items are rated regarding avoidance of the situation. Each item is rated on a four-item Likert scale ranging from 0 (no fear/never avoidance) to 3 (high fear/usually avoidance), with lower scores indicating a better outcome

SECONDARY OUTCOMES:
The secondary outcome is change in Social Cognitions symptoms | 6-months from baseline
  The secondary outcome will be measured by the Social Cognitions Questionnaire (SCQ). SCQ is a 22-item scale that assesses the most common negative automatic thoughts related to SAD. Each thought is rated in terms of how often it occurred in the last week and how much it is believed. The mean scores for frequency (mean ranges from 1 to 5) and for belief (mean ranges from 0 to 100) are computed separately, with lower scores indicating a better outcome.
The secondary outcome is change in depressive symptoms | 6-months from baseline
  The secondary outcome will be measured by the Patient Health Questionnaire (PHQ-9). PHQ-9 is a scale that will be used for assessing depressive symptoms. This scale contains 9 questions answered on a 4-point Likert scale, with numbers from 0 (not at all) to 3 (nearly every day). A higher score reflects more severe symptoms.
The secondary outcome is change in generalised anxiety symptoms | 6-months from baseline
  GAD-7 is a validated questionnaire commonly used to assess generalized anxiety symptoms and their severity. This scale consists of 7 questions answered on a 4-item Likert scale, with numbers from 0 (not at all) to 3 (nearly every day). A higher score reflects more severe symptoms.
The secondary outcome is change in perceived functional impairment | 6-months from baseline
  WSAS is a five-item scale that measures perceived functional impairment across five domains: work, home management, social leisure activities, private leisure activities, and relationships with others. Each item is rated on a 9-point severity scale ranging from 0 (not at all) to 8 (very severely), based on the degree to which the issue impedes one's ability to perform an activity.
The secondary outcome is change in Social participation and social satisfaction | 6-months from baseline
  Social participation and social satisfaction will be measured with Alden and Taylor's scales. Social participation has 13 items that ask about the frequency of participation in social interactions, events, and conversations in the last month. Each item is rated from 1 (not at all) to 7 (frequently). Social satisfaction has five items that ask about satisfaction with relationships with colleagues, friends, and partners in the last month. Each item is rated from 1 (not satisfied at all) to 7 (very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMAD ARSHED, PhD, Principal Investigator — University of Lahore

IPD SHARING:
Plan to Share IPD: No
The study protocol, statistical plan, and results will be disseminated through publications in peer-reviewed Journals.

REFERENCES:
- [Background] Stein MB, Stein DJ. Social anxiety disorder. Lancet. 2008 Mar 29;371(9618):1115-25. doi: 10.1016/S0140-6736(08)60488-2. PMID 18374843
- [Background] Mayo-Wilson E, Dias S, Mavranezouli I, Kew K, Clark DM, Ades AE, Pilling S. Psychological and pharmacological interventions for social anxiety disorder in adults: a systematic review and network meta-analysis. Lancet Psychiatry. 2014 Oct;1(5):368-76. doi: 10.1016/S2215-0366(14)70329-3. Epub 2014 Oct 7. PMID 26361000
- [Background] McHugh RK, Whitton SW, Peckham AD, Welge JA, Otto MW. Patient preference for psychological vs pharmacologic treatment of psychiatric disorders: a meta-analytic review. J Clin Psychiatry. 2013 Jun;74(6):595-602. doi: 10.4088/JCP.12r07757. PMID 23842011
- [Background] Iacobucci G. NICE recommends online therapies to treat depression and anxiety in adults. BMJ. 2023 Mar 1;380:495. doi: 10.1136/bmj.p495. No abstract available. PMID 36858454
- [Background] Thew GR, Kwok APL, Lissillour Chan MH, Powell CLYM, Wild J, Leung PWL, Clark DM. Internet-delivered cognitive therapy for social anxiety disorder in Hong Kong: A randomized controlled trial. Internet Interv. 2022 Apr 18;28:100539. doi: 10.1016/j.invent.2022.100539. eCollection 2022 Apr. PMID 35493437
- [Background] Yoshinaga N, Thew GR, Kobori O, Hayashi Y, Clark DM. Lost in translation? Cultural adaptation of treatment content for Japanese internet-based cognitive therapy for social anxiety disorder. J Behav Cogn Ther. 2021;31(4):363-8. https://doi.org/10.1016/j.jbct.2021.05.004.
- [Background] Brown TA, Barlow DH. Anxiety and Related Disorders Interview Schedule for DSM-5 (ADIS-5)-adult and lifetime version: Clinician manual. Oxford: Oxford University Press; 2014.